CLINICAL TRIAL: NCT00740662
Title: Prospective Study for the Quantification of a Compensatory Increase in Small Bowel Length After Roux-en-Y Gastric Bypass in Morbid Obese Patients by Pre- and Postoperative Length-Measuring With MRI Compared to Intraoperative Length-Measuring
Brief Title: Intraoperative Measuring of Small Bowel Length Compared to Measuring by Magnetic Resonance Imaging (MRI) in Morbid Obese Patients
Status: Terminated | Type: Observational
Why Stopped: Recruiting problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Jean-Marc Heinicke, MD, Department of Visceral and Transplantsurgery, Bern University Hospital
Other Study IDs: KEK248_07
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Morbid Obesity; Weight Loss
Keywords: morbid obesity; small bowel; gastric bypass; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Distal gastric bypass
  Interventions: Procedure: Distal gastric bypass

INTERVENTIONS:
Procedure: Distal gastric bypass — Distal gastric bypass

SUMMARY:
An important step during a gastric bypass operation for the treatment of morbid obesity is the measuring of the small bowel length. At several reoperations we found a length increase of the lowest part of the small intestine of up to 80% compared to the measured length at the initial operation. On the one hand, this reflects a normal technical error of small bowel measuring due to the variable state of contraction of the bowel, but on the other hand, it could also be due to a compensatory increase in intestinal length after the operation. New protocols allow measuring of the small bowel length by MRI. Comparing the preoperative and later on several postoperative measurements by MRI with the initial intraoperative length measuring should allow to validate the new MRI protocol and in the same time quantify the eventual small bowel length increase. We plan to include 20 patients in this study.

DETAILED DESCRIPTION:
Background:

An important step during a gastric bypass operation for the treatment of morbid obesity is the measuring of the small bowel length in order to define the lengths of the alimentary, biliopancreatic and common channel. The measuring itself is technically simple but has always an error due to the variable state of contraction of the small bowel. In distal gastric bypass a common channel length of 100 to 150 cm is chosen which induces an iatrogenic short bowel syndrome. At several reoperations we found a length increase of the common channel of up to 80% compared to the measured length at the initial operation. Former studies seem to indicate that an adaptation of small bowel length may occur in animals with short bowel syndrome or after intestinal bypass surgery. Longterm results of gastric bypass surgery often show weight regain after 3 to 5 years which could be due to the afore mentioned compensatory mechanism.

Newer MRI protocols allow for non-invasive measurement of the small bowel length. Comparing the preoperative and later on several postoperative measurements by MRI with the initial intraoperative length measuring should allow to validate the new MRI protocol and in the same time quantify the eventual small bowel length increase.

Objective:

In-vivo verification of small bowel length measurements made by MRI, quantification of a possible increase of the common channel length in the long run after distal gastric bypass.

Methods:

The preoperative small bowel length measurement by MRI is compared to the length measured intraoperatively. MRIs before discharge postoperatively as well as after 6 and 12 months are used to detect an eventual increase of the common channel length.

ELIGIBILITY:
Inclusion Criteria:

* morbid obese patient
* scheduled for distal gastric bypass
* informed consent for operation and study obtained

Exclusion Criteria:

* history of former small bowel resection
* weight > 150 kg
* history of claustrophobia
* general contraindications for MRI (pacer, joint prosthesis, ear implant, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbid obese patients scheduled for distal gastric bypass
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Small bowel length in vivo compared to measurements by MRI | preoperative, previous to hospital discharge, 6 and 12 months postoperative

SECONDARY OUTCOMES:
Compensatory increase of the common channel (small bowel) after distal bypass | 12 months postoperative
Correlation of longterm weight regain with increase of common channel length | 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Heinicke, MD, Study Director — Department of Visceral and Transplant Surgery, Bern University Hospital; Philipp C Nett, Dr, Principal Investigator — DRNN, Inselspital, Bern University Hospital, Switzerland
Locations (2):
- Switzerland (2):
  - Department of Visceral and Transplantsurgery, Bern University Hopsital, Bern
  - Institute of diagnostic, interventional and pediatric Radiology, Bern University Hospital, Bern

REFERENCES:
- [Background] Miskowiak J, Andersen B. Intestinal adaptation after jejunoileal bypass for morbid obesity: a possible explanation for inadequate weight loss. Br J Surg. 1983 Jan;70(1):27-8. doi: 10.1002/bjs.1800700110. PMID 6824877
- [Background] Swaniker F, Guo W, Fonkalsrud EW, Brown T, Newman L, Ament M. Adaptation of rabbit small intestinal brush-border membrane enzymes after extensive bowel resection. J Pediatr Surg. 1995 Jul;30(7):1000-2; discussion 1003. doi: 10.1016/0022-3468(95)90329-1. PMID 7472920
- [Background] Hughes CA, Ducker DA. Adaptation of the small intestine--does it occur in man? Scand J Gastroenterol Suppl. 1982;74:149-58. PMID 6815778
- [Background] Wyss M, Froehlich JM, Patak MA, Juli CF, Scheidegger MB, Zollikofer CL, Wentz KU. Gradient-enhanced volume rendering: an image processing strategy to facilitate whole small bowel imaging with MRI. Eur Radiol. 2007 Apr;17(4):1081-8. doi: 10.1007/s00330-006-0472-2. Epub 2006 Oct 5. PMID 17021699
- [Background] Patak MA, Froehlich JM, von Weymarn C, Breitenstein S, Zollikofer CL, Wentz KU. Non-invasive measurement of small-bowel motility by MRI after abdominal surgery. Gut. 2007 Jul;56(7):1023-5. doi: 10.1136/gut.2007.120816. No abstract available. PMID 17566036